CLINICAL TRIAL: NCT02477956
Title: Impact of Monthly High Dose Oral Cholecalciferol on Serum 25 Hydroxy Vitamin D Levels in Bariatric Surgery Subjects
Brief Title: Effect of a Monthly High Dose of Vitamin D3 on Bariatric Surgery Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Highly dose of vitamin D3
Record Dates: First submitted 2014-05-12; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Morbid Obesity; Vitamin D Deficiency
Keywords: vitamin D; obesity; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Vitamin D Deficiency; Obesity | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 (Experimental): subjects taking the standard vitamin D protocol with added monthly high dose cholecalciferol of 100,000 IU cholecalciferol
  Interventions: Dietary Supplement: vitamin D3 (Replesta)
- Control (Active Comparator): group of subjects taking the standard vitamin D
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D3 (Replesta) — vitamin D group receive 2 replesta tablets (100,000 IU/month) of cholecalciferol.
  Other Names: Replesta
  Arms: vitamin D3
Dietary Supplement: vitamin D
  Arms: Control

SUMMARY:
Bariatric surgery patients tend to have malabsorption of many micronutrients such as B12, Iron and vitamin D postoperative. So in this study, a monthly high dose of vitamin D3 is giving to patients with their routine supplements and followed up for 6 months.

Hypothesis:Bariatric surgery subjects taking monthly high dose cholecalciferol supplements in addition to the standard vitamin D protocol will have a significant rise in serum vitamin D levels compared to the subjects taking only the usual vitamin D protocol.

DETAILED DESCRIPTION:
Sun exposure and supplement use questionnaire:

A registered dietitian asked each subject for information on sun exposure, vitamins, medications, and any other supplement usage before each blood sample was taken.

Lab analysis included serum hydroxy vitamin D levels pre and 3 months postoperative.

Descriptive statistics which include both the means and standard deviations were calculated on the study variables. A paired sample t-test was used to determine if there was a significant difference in mean values pre and post vitamin D supplementation. An independent sample t-test was used to assess for significant differences in group (control vs. vitamin D supplement) means. A p-value < 0.05 was considered statistically significant. Statistical analyses were done using SPSS Version 21 (SPSS, Chicago, III, USA).

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese and eligible for bariatric surgery

Exclusion Criteria:

* under 18 and over 60 years of age
* elevated serum vitamin D and calcium
* pregnant and lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Impact of monthly high dose oral cholecalciferol on serum 25 hydroxy vitamin D levels in bariatric surgery subjects | one year
  To determine if there is a significant difference in mean serum vitamin D levels in the group of subjects taking the standard vitamin D protocol compared to subjects taking the standard vitamin D protocol with added monthly high dose cholecalciferol after bariatric surgery. This outcome measure is done by analysis of serum 25-OH vitamin D levels.

CONTACTS AND LOCATIONS:
Overall Officials: David Syn, MD, Principal Investigator — Texas Tech University Health Sciences Center; Mallory Boylan, PhD, Study Director — Texas Tech University; Hadil Subih, PhD, Study Chair — Texas Tech University; Shannon Owens, PhD, Study Chair — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States